CLINICAL TRIAL: NCT06281093
Title: Radiofrequency Fields in Neonatology: Exposure and Impact on the Nervous System
Acronym: CHARLINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Brest (Other); Hospices Civils de Lyon (Other); University Hospital, Strasbourg, France (Other); University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2022_843_0089
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Preterm Newborn
Keywords: preterm newborn; radiofrequencies; central and peripheral nervous systems
MeSH Terms: interventions — epicatechin gallate; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionary — Parental questionnaire on pregnancy history and environmental exposure
Other: Daily continuous recording of radiofrequency exposure levels — Daily continuous recording of radiofrequency exposure levels (1 week) by positioning a dosimeter close to the incubator
Other: Follow-up of daily infants clinical parameters — Follow-up of daily infants clinical parameters
Other: recording of cerebral (EEG) — recording of cerebral (EEG)
Other: autonomic nervous (ECG) activity — autonomic nervous (ECG) activity

SUMMARY:
Previously, the investigators showed that preterm newborns are exposed chronically to very low radiofrequency levels in average while hospitalized in NICUs. Most of the infants were nevertheless frequently exposed to transient values above 1 V/m. The investigators also showed that an increase in RF exposure is likely to alter the activity of some neurophysiological functions and their regulatory systems in preterm newborns. The investigators hypothesize that above results are extremely specific to the location of the previous study and may be different in other NICU environments.

This study will aim at quantifying RF levels to which preterm newborns are exposed during their stay in several NICUs spread across the French territory, and assessing its impact on the central and peripheral nervous systems. The first step of this study will be to quantify the precise, continuous and individual levels of daily RF exposure to which each recruited neonate is subjected during his stay in the different NICUs from birth to 1 week postnatal life. Infants' clinical data (medical history, nutrition, morphology...) will also be continually monitored. At 1 week postnatal life, the investigators will investigate cerebral activity (EEG) and autonomic nervous system activity (ECG, heart rate variability). The impact of RF will be evaluated by analyses of the relationship between exposure levels and the various parameters extracted from the neurophysiological investigation phase.

ELIGIBILITY:
Inclusion Criteria:

* preterm newborns born between 26-34 weeks of gestational age

Exclusion Criteria:

* infants infected,
* suffering from neurological disorders,
* serious heart, respiratory, digestive or metabolic diseases;
* infants born from mothers aged less than 18 years old or deprived of their parental rights

Ages: 1 Day to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Variation of the spectral power in the α band (8-12 Hz) of the EEG | one week
  The spectral power in the α band (8-12 Hz) of the EEG

SECONDARY OUTCOMES:
variation of the spectral power in the delta (δ, 0.5-4 Hz) of the EEG | one week

CONTACTS AND LOCATIONS:
Locations (1):
- Amiens University Hospital, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No